CLINICAL TRIAL: NCT02702427
Title: Phase I/II: Treatment of Adenovirus and Cytomegalovirus Infection Post Human Allogeneic Stem Cell Transplantation With Short-term Expanded Virus-specific T Cells
Brief Title: Virus-specific ImmunoTherapy Following Allogeneic Stem Cell Transplantation
Acronym: VISIT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: unsuccessful recruitment
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudra CT2013-002492-17
Record Dates: First submitted 2016-03-01; First posted 2016-03-08 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cytomegalovirus Infection; Adenovirus Infection
Keywords: viral infections post HSCT, virus-specific T-cells
MeSH Terms: conditions — Cytomegalovirus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM 1 (Experimental): Patients with Adenovirus or CMV infection after HSCT and no reduction of viral disease or stable disease with 10E6 viral copies within 2 weeks of antiviral treatment will receive a single infusion of virus-specific T-Cells
  Interventions: Biological: virus-specific T-Cells

INTERVENTIONS:
Biological: virus-specific T-Cells — infusion

SUMMARY:
Invasive infections with CMV and Adenovirus, not responding to virostatic treatment are treated with virusspecific donor derived or autologous virusspecific T-cells.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) is the only treatment option for several haematological diseases. In spite of substantial progress in this field, viral infections, mainly cytomegalovirus (CMV) and adenovirus (HAdV) in the context of delayed immunoreconstitution remain life threatening complications. Weekly screening of high-risk patients and preemptive virostatic treatment has become a current strategy. Unfortunately, treatment with virostatic drugs is associated with substantial nephro- and myelo-toxicity and of limited effectiveness. Human adenovirus (HAdV) and cytomegalvirus (CMV) disseminated infections are associated with mortality rates of up to 50%-60% despite virostatic treatment.

All HSCT patients at the St. Anna Children's Hospital undergo weekly viral quantitative PCR-screening for HAdV and CMV and weekly PB FACS (Fluorescence Activated Cell Sorter)-Analysis according to the local HSCT-diagnostic SOP (Standard Operating Procedure) from day -7 until day +100 Patients with HAdV or CMV viremia will receive preemptive treatment with either gancyclovir (in case of isolated CMV-viremia) or Cidofovir (in case of HAdV viremia or combined HAdV/CMV infection). In case of increasing viremia ≥ 1log despite antiviral treatment for two weeks or stable with 10E6 viral load and the absence of virus specific T-cells in the recipient, the treating physician will check, if the patient is eligible for seVirus-T-cell infusion (see inclusion criteria).

Study Design: Mononuclear Donor-Cells from peripheral blood (100 ml extra donation) will be cryopreserved at the time-point of HSCT. In case of progredient viremia these cells will be stimulated with interleukin-15 and peptides out of the virus molecule, virusspecific T-Cells are enriched for 2-3 logs-teps and potentially alloreactive cells diluted at the same time. This new approach reduces the risk of graft-versus-host-disease (GvHD) and enables the infusion of virus-specific T-cells also from haploidentical donors.

ELIGIBILITY:
Inclusion Criteria:

* Age at timepoint of HSCT ≤18 years undergoing allogeneic stem cell transplantation
* Presence of HAdV or CMV-specific T-cells in the donor or CMV-specific T-cells in the recipient pre-transplant
* Stable (≥ 10E6) or increasing viremia despite antiviral treatment post HSCT
* Absence of HAdV or CMV -specific T cells post HSCT
* Karnofsky / Lansky score >50%
* Pregnancy excluded
* Informed study participation consent is signed

Exclusion Criteria:

* Infusion of polyclonal or monoclonal T-cell directed antibodies within 28 days before seVirus T-Cell infusion
* Multiple organ failure at screening-timepoint seVirus T-Cell infusion
* History of GvHD Gr III-IV or actual GvHD Gr III-IV
* Pregnancy
* Treatment with granulocyte transfusion within the last 72 hours
* Karnofsky / Lansky score <50%
* Subject is unwilling or unable to comply with the study procedures
* High dose treatment with steroids (≥ 2mg/kg/d, methylprednisone-equivalent)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Non pre-existing Immune System Disorders i.e. Allergic reaction, Anaphylaxis, Cytokine release syndrome or Serum sickness of Grade III-IV of seVirus-T-cell infusion within 48 hours from infusion | 48 hours
  assessment is performed according to CTCAE 4.3 Scale
De novo acute GvHD > Gr II or increase of pre-existing GvHD more than 1 grade from 2 weeks post infusion until 8 weeks post infusion | 8 weeks
  assessment is performed according to Glucksberg Scale, modified for paediatic patients from D. Jacobsohn (publication Blood 2008)
Incidence of graft rejection | 8 weeks

SECONDARY OUTCOMES:
Detection of virus-specific T-cells within 8 weeks after T-cell therapy. Measurement of the viral load following the infusion of seVirus-T-cells | 6 months
Correlation of the presence of virus-specific T-cells with partial reduction (>1 log viral copies /ml blood) or complete clearance of viral load | 8 weeks
Tracking of the infused T-cells by NGS (Next Generation Sequencing) of the TCRs (T-Cell Receptors)-beta rearrangements | 3 months
  PBMCs (isolated from about 10ml of peripheral blood) will be resuspended in TRIzol, a ready to use mixture important for later DNA isolation.
  The samples will undergo DNA isolation using a multiplex TCR-beta PCR approach in combination with NGS of the generated amplicons and detailed bioinformatic interpretation of the generated sequence data.
  Current high-throughput sequencing technologies such as Illumina, (HiSeq) enable the analysis of T-cell receptor repertoires in an unprecedented depth.
  As every T-cell harbours a unique TCR-beta rearrangement, we will be able to track T-cell expansion even on a single cell level.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Matthes, MD, Principal Investigator — St. Anna Kinderkrebsforschung
Locations (1):
- St. Anna Children's Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
not planned yet